CLINICAL TRIAL: NCT02747433
Title: Infusing Robot-Assisted Therapy With Motor Learning Principles: An Active Learning Program for Stroke
Brief Title: Robot-Assisted Therapy and Motor Learning: An Active Learning Program for Stroke
Acronym: ALPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Susan Fasoli, ScD OTR/L, Associate Professor, MGH Institute of Health Professions, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2015P002107
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Stroke
Keywords: robot-assisted therapy; task-oriented training; motor learning; cognitive strategy training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single blind study.
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALPS + Robot-Assisted Therapy (RT) (Active Comparator): Armeo and Amadeo robot-assisted intensive upper extremity therapy 1 hr sessions 3x week for 6 weeks plus ALPS training
  Interventions: Device: Robot-Assisted Therapy (RT)
- ALPS + Robot + Task-Oriented Training (RT-TOT) (Active Comparator): Armeo and Amadeo robot-assisted intensive upper extremity therapy 30 mins, 3x week for 6 weeks plus ALPS training. Task oriented training will be provided for remaining 30 min of each treatment session
  Interventions: Device: Robot & Task-Oriented Training (RT-TOT)

INTERVENTIONS:
Device: Robot-Assisted Therapy (RT) — Highly repetitive robot-assisted therapy for paretic arm with Armeo (1 hr sessions, 3x week for 3 weeks) followed by robot-assisted therapy for hand motions with Amadeo (3x week for 3 weeks). Robot training to be accompanied with ALPS motor learning program directed toward UE self management and transfer of training to daily activities in home & community.
  Arms: ALPS + Robot-Assisted Therapy (RT)
Device: Robot & Task-Oriented Training (RT-TOT) — Highly repetitive robot-assisted therapy for paretic arm with Armeo (30 min sessions, 3x week for 3 weeks) followed by robot-assisted therapy for hand motions with Amadeo (3x week for 3 weeks). Task oriented training will be delivered for remaining 30 mins of each treatment session. Robot and task oriented training to be accompanied with ALPS motor learning program directed toward UE self management and transfer of training to daily activities in home & community.
  Arms: ALPS + Robot + Task-Oriented Training (RT-TOT)

SUMMARY:
Stroke is the leading cause of long-term disability in older adults in the United States. At six months after stroke, up to 65% of the more than 795,000 persons who experience a stroke each year continue to have motor impairments that inhibit functional use of the weaker arm during daily activities and negatively impact quality of life. Rehabilitation robots provide clinicians with new treatment options to improve movement and arm function after stroke. The purpose of this pilot study is to develop and test a therapy called the "Active Learning Program for Stroke" (ALPS). We are combining this therapy program with robot-assisted therapy and a home program for the stroke-affected arm and hand.

DETAILED DESCRIPTION:
Little is known about how individuals learn to utilize robot-trained movements during upper extremity (UE) activities in the home and community and whether specific instruction can enhance motor learning and carry-over.. Systematic reviews of robot-assisted therapy for the paretic UE confirm gains in motor capacity as measured by clinical assessments, but provide little evidence of improved UE performance during daily tasks and occupations. These findings may be attributed to the limited availability of rehabilitation robots to train the paretic hand and a primary focus on intensity of practice with little regard for other principles of motor learning and experience-dependent neuroplasticity. These principles, including the salience of training tasks, transfer of acquired skills to similar activities, and active engagement and problem solving, are key to task-oriented training paradigms in stroke (e.g. constraint-induced movement therapy) but have not been well integrated into robot-assisted therapy protocols. The transfer of robot-trained movements to UE activities within the home and community needs further exploration before widespread use in rehabilitation practice is expected.

ELIGIBILITY:
Inclusion Criteria:

* Moderate UE hemiparesis (i.e. some ability to move shoulder, elbow & hand and initial score on the Fugl-Meyer Assessment (FMA) between 21-50/66))
* Intact cognitive function to understand and actively engage in the ALPS robotic therapy procedures (Montreal Cognitive Assessment Score >/=26/30)12 during initial evaluation visit

Exclusion Criteria:

* No more than moderate impairments in paretic UE sensation, passive range of motion, and pain that would limit ability to engage in therapy
* Increased muscle tone as indicated by score of >/= 3 on the Modified Ashworth Scale;
* Hemispatial neglect or visual field loss measured by the symbol cancellation subtest on the Cognitive Linguistic Quick Test 13
* Aphasia sufficient to limit comprehension and completion of the treatment protocol
* Currently enrolled or has plans to enroll in other upper limb therapy/research during the study period
* Contraindications for robot-assisted therapy including recent fracture or skin lesion of paretic UE

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Fasoli, ScD, Principal Investigator — MGH Institute of Health Professions & Spaulding Rehabilitation Hospital; Paolo Bonato, PhD, Study Chair — Spaulding Rehabilitation Hospital & Harvard Medical School
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adans-Dester C, Fasoli SE, Fabara E, Menard N, Fox AB, Severini G, Bonato P. Can kinematic parameters of 3D reach-to-target movements be used as a proxy for clinical outcome measures in chronic stroke rehabilitation? An exploratory study. J Neuroeng Rehabil. 2020 Aug 8;17(1):106. doi: 10.1186/s12984-020-00730-1. PMID 32771020

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the eleven individuals enrolled, one did not meet inclusion criteria and ten were randomized to treatment.
Groups:
- ALPS + Robot-Assisted Therapy (RT): Robot training was combined with the Active Learning Program for Stroke (ALPS) motor learning program directed toward UE self-management and transfer of training to daily activities in home & community.
  Robot-assisted Therapy (RT): Highly repetitive robot-assisted therapy for paretic arm with Armeo (1 hr sessions, 3x week for 3 weeks) followed by robot-assisted therapy for hand motions with Amadeo (1 hr sessions, 3x week for 3 weeks).
- ALPS + Robot + Task-Oriented Training (RT-TOT): Robot and task-oriented training was combined with the Active Learning Program for Stroke (ALPS) motor learning program directed toward UE self-management and transfer of training to daily activities in home & community.
  Robot & Task-Oriented Training (RT-TOT): Highly repetitive robot-assisted therapy for paretic arm with Armeo (30 min sessions, 3x week for 3 weeks) followed by robot-assisted therapy for hand motions with Amadeo (3x week for 3 weeks). Task oriented training was delivered for remaining 30 mins of each treatment session.
Period: Overall Study
Arm/Group | ALPS + Robot-Assisted Therapy (RT) | ALPS + Robot + Task-Oriented Training (RT-TOT)
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALPS + Robot-Assisted Therapy (RT) | ALPS + Robot + Task-Oriented Training (RT-TOT) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (19.8) | 46.5 (19.5) | 53.2 (19.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Fugl-Meyer Assessment-Upper Extremity [Mean (Standard Deviation); unit: units on a scale] | 30.4 (6.7) | 34.0 (12.4) | 32.2 (9.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fugl-Meyer Assessment (FMA) - Upper Extremity Subtest
Description: The FMA will examine changes in motor function, pain and sensation in the paretic UE between baseline, post-intervention and 1-month follow-up assessments. The FMA upper extremity subtest contains 33 items, scored as 0= unable, 1=partial ability, 2= faultless with a total possible score of 66 points. Change was calculated as the value at the 1 month follow-up assessment minus the value at baseline to reflect retention of motor function following intervention.
Time Frame: Baseline and 1-month follow-up
Population: Primary aims were to examine the feasibility and effects of the Active Learning Program for Stroke (ALPS) on paretic upper extremity function when combined with either robot-assisted therapy or robot-assisted therapy plus task-oriented training. In the 3rd Arm, data from both groups were combined to examine effects of ALPS + intensive UE training.
Measure: Median (Full Range); unit: score on a scale
Groups:
- ALPS + RT + RT-TOT: Participants in both groups received the Active Learning Program for Stroke (ALPS) motor learning program directed toward upper extremity (UE) self-management and transfer of robot-trained UE skills to daily activities in the home & community.
  The ALPS protocol was administered to individuals in the RT group who received intensive upper extremity robot-assisted therapy with the Armeo and Amadeo robots, 1 hr sessions 3x week over 6 weeks (ALPS + RT) and to individuals who received robot-assisted therapy and task- oriented training during each session (ALPS + RT-TOT). Individuals in the RT-TOT group received robot-assisted therapy with the Armeo and Amadeo robots for 30 mins plus task-oriented training for the remaining 30 min of each treatment session, 3x week for 6 weeks.
Arm/Group | ALPS + Robot-Assisted Therapy (RT) | ALPS + Robot + Task-Oriented Training (RT-TOT) | ALPS + RT + RT-TOT
Number analyzed (Participants) | 5 | 5 | 10
score on a scale | 11.0 [9.0 to 14.0] | 2.0 [-1.0 to 8.0] | 8.5 [-1.0 to 14.0]

2. Primary Outcome: Change From Baseline in Wolf Motor Function Test (WMFT)
Description: The WMFT examined changes in ability to complete timed, functionally-based activities with the paretic UE between baseline, post-intervention and 1-month follow-up assessments. The task rate was calculated as the average # of times that each test item could be completed within 1 minute. Here we report the change in task rate scores between admission and 1 month follow-up assessments to reflect retention of motor function following intervention. A higher number indicates improved task completion.
Time Frame: Baseline and 1-month follow-up
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | ALPS + Robot-Assisted Therapy (RT) | ALPS + Robot + Task-Oriented Training (RT-TOT) | ALPS + RT + RT-TOT
Number analyzed (Participants) | 5 | 5 | 10
units on a scale | 10.22 [-1.18 to 10.77] | 3.07 [-0.52 to 8.47] | 6.98 [-1.18 to 10.77]

3. Primary Outcome: Change From Baseline on Confidence in Arm and Hand Movement (CAHM) Scale
Description: The CAHM is a self-report assessment in which participants are asked to rate their confidence (0-100%) in successfully using their paretic UE for a variety of everyday activities. Change in confidence ratings between baseline, post-intervention and 1-month follow up assessments were examined. A higher score indicates greater confidence. We report change scores between admission and 1 month follow up assessments to reflect retention of scores following intervention.
Time Frame: Baseline and 1-month follow-up
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ALPS + Robot-Assisted Therapy (RT) | ALPS + Robot + Task-Oriented Training (RT-TOT) | ALPS + RT + RT-TOT
Number analyzed (Participants) | 5 | 5 | 10
score on a scale | 8.00 [-14.00 to 21.75] | 9.50 [4.25 to 49.00] | 8.75 [-14.00 to 49.00]

4. Secondary Outcome: Change From Baseline on Motor Activity Log (MAL) - Amount of Use (AOU) Scale
Description: The MAL has been widely used in stroke rehabilitation studies to measure self-reported amount and quality of paretic arm use during daily activities. Participant's self-reported amount of use (AOU) and how well the task was performed (HW) are rated on a scale from 0=not used at all to 5=as much or as well as before the stroke. Higher scores indicate greater perceived motor function in the paretic arm & hand.
  We report change scores in amount of use (AOU) between admission and 1 month follow up assessments to reflect retention of motor function following intervention..
Time Frame: Baseline and 1-month follow-up
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | ALPS + Robot-Assisted Therapy (RT) | ALPS + Robot + Task-Oriented Training (RT-TOT) | ALPS + RT + RT-TOT
Number analyzed (Participants) | 5 | 5 | 10
units on a scale | 0.89 [0.12 to 1.75] | 0.52 [0.15 to 0.83] | 0.59 [0.12 to 1.75]

5. Secondary Outcome: Change From Baseline on Motor Activity Log (MAL) - How Well (HW) Scale
Description: The MAL has been widely used in stroke rehabilitation studies to measure self-reported amount and quality of paretic arm use during daily activities. Participant's self-reported amount of use (AOU) and how well the task was performed (HW) are rated on a scale from 0=not used at all to 5=as much or as well as before the stroke. Higher scores indicate greater perceived motor function in the paretic arm & hand.
  We report change scores in how well the function was performed between admission and 1 month follow up assessments to reflect retention of motor function following intervention..
Time Frame: Baseline and 1-month follow-up
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Groups:
- ALPS + Robot & Task-Oriented Training (RT-TOT): Robot and task-oriented training was combined with the Active Learning Program for Stroke (ALPS) motor learning program directed toward UE self-management and transfer of training to daily activities in home & community.
  Robot & Task-Oriented Training (RT-TOT): Highly repetitive robot-assisted therapy for paretic arm with Armeo (30 min sessions, 3x week for 3 weeks) followed by robot-assisted therapy for hand motions with Amadeo (3x week for 3 weeks). Task oriented training was delivered for remaining 30 mins of each treatment session.
Arm/Group | ALPS + Robot-Assisted Therapy (RT) | ALPS + Robot & Task-Oriented Training (RT-TOT) | ALPS + RT + RT-TOT
Number analyzed (Participants) | 5 | 5 | 10
units on a scale | 1.00 [0.06 to 1.55] | 0.71 [0.27 to 0.93] | 0.81 [0.06 to 1.55]

6. Secondary Outcome: Change From Baseline on Modified Ashworth Scale (MAS)
Description: The MAS examined changes in muscle tone in the paretic UE . Scores range from 0=no increase in muscle tone to 4=affected part(s) rigid in flexion or extension. Tested muscle groups include shoulder internal rotators, elbow flexors/extensors, supinators, pronators, wrist flexors/extensors, finger flexors/extensors. Lower scores indicate better motor function. We present the change scores between admission and 1 month follow up assessments to reflect retention of motor function following intervention. .
Time Frame: Baseline and 1-month follow-up
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | ALPS + Robot-Assisted Therapy (RT) | ALPS + Robot & Task-Oriented Training (RT-TOT) | ALPS + RT + RT-TOT
Number analyzed (Participants) | 5 | 5 | 10
units on a scale | 0.00 [-0.22 to 0.22] | 0.22 [-0.22 to 0.39] | 0.03 [-0.22 to 0.39]

7. Secondary Outcome: Change From Baseline on Stroke Impact Scale (SIS) - Hand Domain
Description: The SIS measured changes in activity and participation due to stroke. The SIS assesses eight domains including strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion, memory & thinking, and participation/role function. A transformed score for each domain is calculated from its raw score and represented by a 100 point scale, with higher scores representing better performance. We report the change in transformed scores for the hand function domain, between admission and 1 month follow up assessments to reflect retention of motor function following intervention.
Time Frame: Baseline and 1-month follow-up
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ALPS + Robot-Assisted Therapy (RT) | ALPS + Robot & Task-Oriented Training (RT-TOT) | ALPS + RT + RT-TOT
Number analyzed (Participants) | 5 | 5 | 10
score on a scale | 8.00 [0.00 to 24.00] | 4.00 [4.00 to 20.00] | 4.00 [0.00 to 24.00]

8. Secondary Outcome: Change From Baseline on Stroke Impact Scale (SIS) - Percent Recovery
Description: The SIS measures changes in activity and participation due to stroke. The SIS assesses eight domains including strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion, memory & thinking, and participation/role function. A transformed score for each domain is calculated from its raw score and represented by a 100 point scale, with higher scores representing better performance. We report the participants' rating of stroke recovery (how much the participant feels that he/she has recovered from stroke with 0=no recovery, 100=full recovery), between admission and 1 month follow up assessments to reflect retention of motor function following intervention.
Time Frame: Baseline and 1-month follow-up
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ALPS + Robot-Assisted Therapy (RT) | ALPS + Robot & Task-Oriented Training (RT-TOT) | ALPS + RT + RT-TOT
Number analyzed (Participants) | 5 | 5 | 10
score on a scale | 20.00 [-20.000 to 25.00] | 5.00 [-6.00 to 10.00] | 10.00 [-20.00 to 25.00]

9. Secondary Outcome: Change From Baseline in Movement Time During Reach-to-Target Task
Description: Participants were asked to reach forward from a designated starting position toward a panel with 12 numbered targets positioned in a clockwise-fashion 20 cm from from its center. The center of the target was aligned with the acromion of the paretic arm and reflective markers were attached to locations on the trunk and paretic arm to allow recording of kinematic data via 3-D motion capture (Vicon Motion Systems Ltd. UK) for off-line analysis. Data from reaching movements to all targets were combined for analysis. We report the median values for Movement Time (sec) for the entire sample at the time of a discharge assessment immediately following the 6-week intervention.
Time Frame: Baseline and immediately after 6-week intervention
Population: Because the primary aim of this pilot was to explore the combined effects of the Active Learning Program for Stroke (ALPS ) and robot-assisted therapy/task oriented training, a decision was made a priori that this data would be collected and analyzed in a pooled manner for this exploratory endpoint.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | ALPS + RT + RT-TOT
Number analyzed (Participants) | 10
seconds
  Baseline | 2.37 [1.95 to 2.86]
  Discharge | 2.17 [1.94 to 2.51]

10. Secondary Outcome: Change From Baseline in Log Dimensionless Jerk During Reach-to-Target Task
Description: Participants were asked to reach forward from a designated starting position toward a panel with 12 numbered targets positioned in a clockwise-fashion 20 cm from from its center. The center of the target was aligned with the acromion of the paretic arm and reflective markers were attached to locations on the trunk and paretic arm to allow recording of kinematic data via 3-D motion capture (Vicon Motion Systems Ltd. UK) for off-line analysis. Data from reaching movements to all targets were combined for analysis. We report the median values for Log Normalized Jerk, a measure of movement smoothness during reach, for the entire sample at the time of a discharge assessment immediately following the 6-week intervention.
Time Frame: Baseline and immediately after 6-week intervention
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: dimensionless
Arm/Group | ALPS + RT + RT-TOT
Number analyzed (Participants) | 10
dimensionless
  Baseline | -18.89 [-19.66 to -18.25]
  Discharge | -18.14 [-19.21 to -17.97]

ADVERSE EVENTS:
Time Frame: Adverse event data for participants was collected during a 12 week period ranging from baseline to one-month follow-up assessments.
Groups:
- Robot-Assisted Therapy (RT): Armeo and Amadeo robot-assisted intensive upper extremity therapy 1 hr sessions 3x week for 6 weeks plus ALPS training
  Robot-Assisted Therapy (RT): Highly repetitive robot-assisted therapy for paretic arm with Armeo (1 hr sessions, 3x week for 3 weeks) followed by robot-assisted therapy for hand motions with Amadeo (3x week for 3 weeks). Robot training was accompanied with ALPS motor learning program directed toward UE self management and transfer of training to daily activities in home & community.
- Robot & Task-Oriented Training (RT-TOT): Armeo and Amadeo robot-assisted intensive upper extremity therapy 30 mins, 3x week for 6 weeks plus ALPS training. Task oriented training was provided for remaining 30 min of each treatment session
  Robot & Task-Oriented Training (RT-TOT): Highly repetitive robot-assisted therapy for paretic arm with Armeo (30 min sessions, 3x week for 3 weeks) followed by robot-assisted therapy for hand motions with Amadeo (3x week for 3 weeks). Task oriented training was delivered for remaining 30 mins of each treatment session. Robot and task oriented training was accompanied with ALPS motor learning program directed toward UE self management and transfer of training to daily activities in home & community.
Arm/Group | Robot-Assisted Therapy (RT) | Robot & Task-Oriented Training (RT-TOT)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
We are unable to report results of accelerometer data due to technical problems.Surface electromyography (EMG) during reach-to-target kinematic assessment was collected for a separate study by Dr. Bonato and has not been analyzed by co-investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT02747433/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT02747433/ICF_001.pdf